CLINICAL TRIAL: NCT04673266
Title: Romiplostim for Prevention of Severe Chemotherapy Induced Thrombocytopenia in Lymphoma Patients - Phase II Study
Brief Title: Using Romiplostim to Treat Low Platelet Counts During Chemotherapy in People With Lymphoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Amgen (Industry); Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20-492
Record Dates: First submitted 2020-12-14; First posted 2020-12-17 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Lymphoma Patients; Thrombocytopenia
Keywords: Romiplostim; 20-492
MeSH Terms: conditions — Thrombocytopenia | interventions — romiplostim

STUDY DESIGN:
Intervention Model Description: A single-center, open-label phase II study.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- romiplostim (Experimental): Romiplostim will be administered from the beginning of the next chemotherapy cycle with a starting dose of 3 mcg/kg subcutaneously. Dose will be titrated based on nadir of the platelet counts during the prior cycle. The maximum dose of romiplostim will be 6 mcg/kg.
  Interventions: Drug: Romiplostim

INTERVENTIONS:
Drug: Romiplostim — All patients will begin weekly (+/- 2 days) romiplostim at 3 mcg/kg subcutaneously. The romiplostim dose will be titrated, based on weekly CBC/platelet counts.

SUMMARY:
The purpose of this study is to see if the study drug, romiplostim, helps low platelet count caused by standard chemotherapy treatment for lymphoma. This study will also look at whether romiplostim can prevent the need for chemotherapy dose delays, chemotherapy dose reductions, and platelet transfusions. In addition, we will determine how safe it is to give romiplostim to people with lymphoma who have low platelet count from chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients ≥ 18 years old diagnosed with any type of lymphoma.
* Receiving chemotherapy-based treatment known to cause thrombocytopenia. Eligibility is limited to regimens with a 21-day cycle. Previous single-agent anti-CD20 antibody or radiotherapy will not count as a line of treatment. Eligible regimens include those based on a platinum backbone (e.g. ICE, DHAX, DHAP, GemOx, GDP, ESHAP), those based on a doxorubicin backbone (e.g. CHOP, CDOP, HyperCVAD, BEACOPP) or on a high-dose cytarabine backbone (e.g.HiDAC). Of note, treatment programs which involve sequential administration of two or more regimens (e.g. CHOP->ICE or CHOP-DHAX) are eligible as long as the patient is planned for at least two more cycles of the regimen on which the CIT was initially observed. Regimens with inherent dose-adjustments by blood counts (e.g. da-EPOCH) are ineligible unless the treating oncologist is not planning to increase treatment doses on subsequent cycles.
* History of a severe treatment-related thrombocytopenia during the most recent cycle of treatment, as defined by one or more of the following criteria:

  * PLT < 50,000 on day 1 (- 2 days) of the subsequent treatment cycle.
  * Grade 4 thrombocytopenia, defined as PLT <25,000 cells/mcl and/or transfusion for thrombocytopenia or bleeding. Need for PLT transfusion in order to meet minimal PLT criteria for invasive procedures will not count for eligibility.
* Patient is planned for at least one more cycle of chemotherapy.
* ECOG Performance Status of ≤ 2 (Karnofsky ≥50%, see Appendix A - ECOG/Karnofsky performance status scale).
* Patients must have normal organ function as defined below on day 1 of the prior cycle:

  * Absolute neutrophil count ≥ 1,000/mcL - use of gCSF is acceptable for eligibility
  * Hemoglobin ≥ 7 g/dL - transfusion support is acceptable for eligibility
  * Total bilirubin ≤ 3x the institutional ULN
  * AST and ALT ≤ 3x institutional upper limit of normal
* Human immunodeficiency virus (HIV)-infected patients on effective antiretroviral therapy with undetectable viral load are eligible for this trial, provided there are no anticipated interactions between antiretroviral treatment and the study drug.
* Women of child-bearing potential (WOCBP) and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation.
* Ability to understand and the willingness to sign a written informed consent document prior to participation in the study and any related procedures being performed. Legally Authorized Representatives are permitted.

Exclusion Criteria:

* History of or concurrent hematological malignancy other than lymphoma (acute or chronic leukemia, myelodysplastic syndrome [MDS], myeloproliferative neoplasm, multiple myeloma). Patient with composite/concurrent lymphoma or Richter's transformation are eligible.
* History of allogeneic hematopoietic stem cell transplantation (SCT). Patients with a prior autologous SCT or CAR-T treatment are eligible.
* Patients with history of symptomatic venous thrombotic event (VTE), such as deep vein thrombosis (DVT) or pulmonary embolism (PE) who is unable to tolerate anticoagulation. Patients who have completed their indicated course of anticoagulation prior to enrollment or are tolerating ongoing anticoagulation are eligible. Patients with VTE associated with central venous catheter are eligible.
* Patients with history of symptomatic arterial thrombotic events such as myocardial infarction, ischemia cerebral vascular accident, or transient ischemic attack within 4 months prior to enrollment.
* Patients who have thrombocytopenia related to pre-existing ITP.
* Major surgery within 26 days prior to enrollment, or minor surgery within 3 days prior to enrollment.
* Solid-tumor malignancy metastatic or locally-advanced unresectable within the last 5 years that could adversely affect subject safety or longevity, create the potential for drug-drug interactions, or compromise the interpretation of study results.
* Concurrent therapy with other investigational agents.
* Within 4 months prior to enrollment, any history of active congestive heart failure (New York Heart Association [NYHA] Class III to IV), symptomatic ischemia, uncontrolled arrhythmias, clinically significant electrocardiogram (ECG) abnormalities, screening ECG with corrected QT (QTc) interval of > 470 msec, pericardial disease, or myocardial infarction.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, renal failure requiring hemodialysis, or psychiatric illness/social situations that would limit compliance with study requirements. These include abnormal laboratory values, that could cause unacceptable safety risks or compromise compliance with the protocol.
* Patients are excluded from this study if pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the trial, starting with the screening visit through 180 days after the last dose of trial treatment.
* Patient has acute viral hepatitis (typically defined by elevated AST/ALT), or a history of chronic or active HBV or HCV infection (HBcAb or HBsAg positive and detectable serum/plasma HBV DNA, or HCV Ab positive and detectable serum/plasma HCV RNA).
* Patients with any significant history of non-compliance to medical regimens or unwilling or unable to comply with the instructions given to him/her by the study staff.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2020-12-14 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
measure of incidence of indication for dose delays | 1 year
  defined as PLT < 50,000 cells/mcl) at the end of cycle 1 (C1D21±2d); presence of grade 4 thrombocytopenia (<25,000 cells/mcl) at any time throughout the treatment cycle; or indication for a PLT transfusion for thrombocytopenia or for bleeding at any time throughout the treatment cycle.

CONTACTS AND LOCATIONS:
Overall Officials: Zachary Epstein-Peterson, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (8):
- United States (8):
  - University of Miami - Sylvester Comprehensive Cancer Center, Miami, Florida
  - Memorial Sloan Kettering Basking Ridge (All Protocol Activites), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (All Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (All Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Commack (All Protocol Activities), Commack, New York
  - Memorial Sloan Kettering Westchester (All Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York
  - Memorial Sloan Kettering Nassau (All Protocol Activities), Uniondale, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm